CLINICAL TRIAL: NCT02737839
Title: Adaptation of the STEPPING ON Fall Prevention Program for Older Adults Receiving Cancer Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201603069
Record Dates: First submitted 2016-03-22; First posted 2016-04-14 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Geriatric Disorder; Cancer; Patient Fall
MeSH Terms: conditions — Neoplasms | interventions — House Calls; Patient Health Questionnaire

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1: STEPPING ON (Experimental): * Adaptation Waves is to adapt Stepping On to the oncology setting/Pilot Waves is to determine the feasibility & acceptability of the program for older adults receiving cancer care/Gait & Balance Waves is to determine whether the participants experience changes in their gait & balance
    * Complete baseline questionnaires about Instrumental Activities of Daily Living, Medical Outcome Study Activities, Karnofsky Performance Status, falls in past 3 months, medications, comorbidities, vision & hearing, The Falls Behavioral Scale, The Falls Efficacy Scale-International, Patient Reported Outcome pain, PRO neuropathy
    * 7 week STEPPING ON program is multi-component learning environment which has shown to help reduce falls
    * A home visit to gather any feedback on the experience of the program
    * Follow-up questionnaires up to 3 months after completion of the program
  * Participants may elect to participate in a "booster session" to reinforce concepts 3-6 months after completion of the program
  Interventions: Other: Stepping On Education Program; Other: Home visit; Other: Patient Questionnaire; Other: Mini-Balance Evaluation Systems Test; Other: GAITRite; Other: Precise measure of movement testing

INTERVENTIONS:
Other: Stepping On Education Program
Other: Home visit
Other: Patient Questionnaire — -Includes questions about demographics, activity level, performance status, falls, medication, comorbidities, hearing, vision, pain, and neuropathy
Other: Mini-Balance Evaluation Systems Test — * The Mini-BESTest includes 14-items that assess balance across four domains: 1) anticipatory postural adjustments, 2) reactive postural responses, 3) sensory orientation, and 4) stability in gait. Each item is rated on a 0-2 scale with 0 indicating poor balance and 2 indicating no impairment. The total possible score on the Mini-BESTest is 28 points
  * Balance testing will take approximately 15 minutes.
  Other Names: Mini-BESTest
Other: GAITRite — * Gait will be assessed using the 4.87-m GAITRite
  * The GAITRite is a computerized mat that allows for measurement of spatiotemporal measures (e.g., gait velocity, stride length) of gait. We will measure gait in the following conditions: 1) comfortable forward, 2) fast-as-possible, and 3) dual-task. For comfortable forward, participants will be asked to walk at their self-perceived normal pace. For fast-as-possible, participants will be asked to walk as quickly and safely as possible. For dual-task, participants will be asked to walk at their comfortable pace forward while saying as many words that begin with a letter given to them just prior to the start of the trial. Participants will complete five trials of each condition. Gait testing will take approximately 15 minutes.
Other: Precise measure of movement testing — We will conduct additional movement-based testing with participants wearing small, portable sensors (APDM, Inc., Portland, OR). These sensors allow for precise measurement of movement characteristics. The sensors will be worn on the outside of clothing and will be placed on the following body locations: 1) sternum, 2) low back, 3) right wrist, 4) left wrist, 5) right ankle, and 6) left ankle. The participants will wear these sensors during the following movement tasks: 1) Two Minute Walk Test, 2) Timed Up & Go, 3) Dual Timed Up & Go, 4) Stand and Walk (SAW), and 5) 360 Degree Turn test. These sensors will allow for capture of precise measures postural sway, arm swing, gait variability, and many other variables the proposed movement tasks.

SUMMARY:
Chronic disease self-management is the ability of the individual, in conjunction with family, community and healthcare professionals to manage symptoms, treatments, lifestyle changes and psychosocial, cultural and spiritual consequences associated with a chronic condition. Self-management strategies have been successfully used in supportive care and survivorship in oncology. Stepping On, a multi-component program using a small-group learning environment, reduces falls by 31%. It empowers participants with knowledge about fall-risk, exercise, medications and environmental hazards to self-manage their risk of falls over 7 weeks of educational sessions, followed by a home visit. The research in this proposal will yield the adaptation of the effective group-education-based fall-prevention intervention Stepping On, tailored to cancer patients, feasible for testing in a multi-institutional trial, and ultimately scalable in the oncology setting.

ELIGIBILITY:
Inclusion Criteria for Patient Participants:

* Age ≥70 years.
* Reports a fall within the past 1 year OR self-reports that they are concerned about falling.
* Receiving systemic cancer therapy (including conventional chemotherapy, novel/targeted agents, immunotherapy, monoclonal antibody therapy, oral tyrosine kinase inhibitors, or hormonal agents) OR will begin systemic therapy within the next 4 weeks.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria for Patient Participants:

* Life expectancy <6 months.
* Unable to understand written or spoken English.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Percent of participants who completed the 7 education sessions | Completion of all participants in the Pilot Wave groups (approximately 85 weeks)
  -The Pilot Waves will only be looked at for this outcome measure

SECONDARY OUTCOMES:
Percent of participants consented among approached potential participants | Completion of accrual (approximately 18 months)
  -The Pilot Waves will only be looked at for this outcome measure
Fall rate during participation | Completion of participation (approximately 20 weeks)
  -The Pilot Waves will only be looked at for this outcome measure
Changes in score in the Falls-Efficacy Scale - International as measured by fear-of-falling | Completion of participation (approximately 20 weeks)
  -The Pilot Waves will only be looked at for this outcome measure
Behavior change intention in preventing falls | Completion of participation (approximately 20 weeks)
  * The Pilot Waves will only be looked at for this outcome measure
  * To measure behavior change intention in preventing falls the participant will be asked 24 questions about how they prevent falls. Answers to choose from include never, sometimes, often, always, or does not apply.
Change in Pain Patient Reported Outcome (PRO) | Completion of participation (approximately 20 weeks)
  -5 questions to ask participant about their pain levels and how the pain interfered with their daily lives, answers range from not at all to very much
Measure changes in balance waves | Baseline and 1 month after completion of participation (approximately 20 weeks)
  -The Gait & Balance Waves will only be looked at for this outcome measure
Measure changes in gait waves | Baseline and 1 month after completion of participation (approximately 20 weeks)
  -The Gait & Balance Waves will only be looked at for this outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Clifton, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu